CLINICAL TRIAL: NCT03588351
Title: Chitosan,Chitosan Nanoparticles,and Chlorhexidine Gluconate, as Intra Canal Medicaments in Primary Teeth: An In-vivo Study
Brief Title: Chitosan,Chitosan Nanoparticles,and Chlorhexidine Gluconate, as Intra Canal Medicaments in Primary Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Abozed, Marwa Ahmed Abozed, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED-3-17
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Necrotic Pulp
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- chlorhexidine gluconate (Active Comparator): GROUP I: - 15 teeth will be treated with specially prepared gel containing chlorhexidine gluconate as intracanal medicament .
  Interventions: Drug: chlorhexidine gluconate
- chitosan nanoparticles gel (Experimental): GROUP II: - 15 teeth will be treated with specially prepared gel containing chitosan nanoparticles that ready to use as intracanal medicament.
  Interventions: Drug: chitosan nanoparticles gel
- chitosan gel (Experimental): Group III: 15teeth will be treated with specially prepared gell containing chitosan that ready to use as intra medicament .
  Interventions: Drug: chitosan gel

INTERVENTIONS:
Drug: chitosan nanoparticles gel — intracanal medicament
  Other Names: CSNPs
  Arms: chitosan nanoparticles gel
Drug: chitosan gel — intracanal medicament
  Other Names: CS
  Arms: chitosan gel
Drug: chlorhexidine gluconate — intracanal medicament
  Other Names: CHX
  Arms: chlorhexidine gluconate

SUMMARY:
Aim of the present study is to assess the in vivo susceptibility of root canal bacteria to Chitosan,Chitosan nanoparticles ,and Chlorhexidine gluconate when used as intra canal medicaments in necrotic primary molars

DETAILED DESCRIPTION:
Primary teeth with necrotic pulp are a common problem in pediatric dentistry especially in very young children before first permanent molar eruption. Early loss of primary teeth can cause a number of problems, including space loss, esthetic, phonetic or functional problems. However, some of the infected primary teeth can remain functional until the exfoliation via endodontic treatment. Pulpectomy is indicated in primary teeth with necrotic pulp in which the radicular tissue exhibits clinical signs of chronic inflammation.

The primary objective of pulp therapy is to maintain the integrity and health of the teeth and their supporting tissues. One of the most important aims of pulpectomy treatment is to eradicate or substantially reduce the microbial load in the root canal system. Currently, insignificant data is available regarding the identification of microbiota in deciduous teeth with pulp necrosis and periapical pathosis. However, documentation exists in relation to the polymicrobial nature of microbes predominated by anaerobes in the root canals of deciduous teeth with necrotic pulp and periapical lesions similar to permanent teeth.

Various microorganisms isolated from infected root canals include Streptococci, Staphylo-coccus, Diptheroids, Peptostreptococcus, Lactoba-cilli, Propionibacterium, Actinomyces, Bacteroides, Fusobacterium etc.

The commonly isolated facultative anaerobes microorganisms from primary root canals, Enterococcus faecalis was isolated in 30% of cases, Escherichia coli in 28.4%, Staphylococcus aureus in 25%, α-hemolytic Streptococci in 15% and Proteus mirabilis in 1.6% of cases.

E. faecalis is a persistent organism that plays a major role in the etiology of persistent periradicular lesions after root canal treatment. It is commonly found in high percentage of root canal failures and is able to survive in the root canal as a single organism or as a major component of the flora.

Therefore, intracanal medication was advocated to further reduce bacteria in the root canal system and reduce the failure of root canal treatment. Thus, chemomechanical debridement using intracanal medicament and irrigants is essential to eliminate these microorganisms, and their by-products that remained in the pulpal space which was inaccessible to systemic antibiotics and root canal instrumentations.

Chlorhexidine (CHX) usually used as a root canal irrigant especially in primary molars owing to its biocompatibility, substantivity and wide antimicrobial activity.

Recently there is an increase interest in using natural product in medical fields. Chitosan is a natural and non-toxic polysaccharide with many biological applications, particularly as an antimicrobial agent. Chitosan nanoparticle is a bioactive and environment friendly material with unique physicochemical properties .

To date, none of the studies has consistently investigated the effects of Chitosan as new alternative when used as root canal medicament in primary teeth. Therefore the present study aimed to compare in vivo susceptibility of root canal bacteria to chitosan, chitosan nanoparticals, and chlorhexidine gluconate as intra canal medicaments in necrotic primary molars.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children.
* Age 4-7 years
* Children should have at least one non vital and restorable mandibular molar .
* Cooperative children.
* Children that did not take any antibiotic for at least one month before sample collection

Exclusion Criteria:

* Medically compromised children.
* Children under antibiotic therapy.
* Non restorable molars.
* Root resorption more then half of the root length.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-15 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
assess the in vivo susceptibility of root canal bacteria to Chitosan,Chitosan nanoparticals ,and Chlorhexidine gluconate when used as intra canal medicaments in necrotic primary molars. | 3 month
  antibacterial effect of Chlorhexidine Gluconate, Chitosan,Chitosan Nanoparticl on necrotic primary tooth

CONTACTS AND LOCATIONS:
Overall Officials: Marwa A Abozed, BDSC, Principal Investigator — Faculty of Dentistry Ain shams University, Cairo, Egypt
Locations (1):
- Ain shames university faculty of dentistry, Cairo, Egypt